CLINICAL TRIAL: NCT07169188
Title: A 12-Week Randomized, Controlled, Single-Blind, Clinical Study Investigating the Efficacy of an Experimental Toothpaste Containing Stannous Fluoride in Improving Gingival Health
Brief Title: A Clinical Study Investigating the Efficacy of an Experimental Toothpaste Containing Stannous Fluoride in Improving Gingival Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 400031
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Dental Plaque; Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Toothpaste (Experimental): Participants will brush their teeth with full ribbon of test toothpaste applied on head of toothbrush provided for one timed minute twice a day (morning and evening) for 12 weeks.
  Interventions: Drug: Test Fluoride Toothpaste
- Reference Toothpaste (Active Comparator): Participants will brush their teeth with full ribbon of reference toothpaste applied on head of toothbrush provided for one timed minute twice a day (morning and evening) for 12 weeks.
  Interventions: Drug: Colgate Cavity Protection Toothpaste

INTERVENTIONS:
Drug: Test Fluoride Toothpaste — Toothpaste containing 0.454% SnF2, 0.3% zinc chloride (ZnCl2) and 1% alumina.
  Arms: Test Toothpaste
Drug: Colgate Cavity Protection Toothpaste — Regular fluoride toothpaste containing 0.76% sodium monofluorophosphate.
  Arms: Reference Toothpaste

SUMMARY:
The aim of this study is to evaluate the ability of an experimental toothpaste, containing 0.454 percent (%) Stannous Fluoride (SnF2) to improve gingival health and reduce plaque accumulation compared to a regular fluoride toothpaste (reference dentifrice) in participants with localized, plaque-induced, gingivitis.

DETAILED DESCRIPTION:
This will be a single-center, 12 weeks, randomized, controlled, examiner-blind, 2 treatment arms, parallel group design clinical study to evaluate the efficacy of an experimental toothpaste containing 0.454% SnF2, used twice daily in reducing gingivitis and plaque accumulation in a population with clinically measurable levels of gingivitis. The clinical efficacy of the experimental toothpaste will be compared with a reference dentifrice, a commercially available, regular fluoride toothpaste. Additionally, unstimulated saliva samples will be collected from a sub-set of the randomized participants pre-brushing and at 15, 30, 60 and 120 minutes post-brushing which will be analyzed for tin concentration to investigate the retention of the stannous [tin (II)] ion within the oral cavity. Approximately 160 participants will be randomized to ensure approximately 144 evaluable participants complete the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided a signed and dated informed consent document indicating that they have been informed of all pertinent aspects of the study before any assessment is performed.
2. Participant is of either biological sex and any gender.
3. Participant is, at the time of screening, aged 18-70 years, inclusive.
4. Participant is willing and able to comply with scheduled visits, treatment plan and all study procedures and Lifestyle Considerations.
5. Participant is in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history or upon oral examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
6. Participant with oral health that meets all the following:

   1. At Visits 1 and 2, has at least 20 natural, permanent teeth (excluding 3rd molars) with at least 40 evaluable surfaces for MGI and TPI assessments.
   2. At Visit 2, has, in the opinion of the examiner, localized plaque-induced gingivitis with 10-30% bleeding sites from the BI assessment and with an overall TPI score >= 1.5.

Exclusion Criteria:

1. Participant is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or a Haleon employee directly involved in the conduct of the study or a member of their immediate family.
2. Participant has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
3. Participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
4. Participant has any other clinical serious or unstable conditions (example, cardiovascular diseases, diabetes, liver disorders, and kidney disorders) which could have affected study outcomes and/or participant safety.
5. Participant is breast feeding or is pregnant (self-reported) or intending to become pregnant over the duration of the study.
6. Participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
7. Participant is unwilling or unable to comply with the Lifestyle Considerations described in this protocol.
8. Participant is a current or ex (stopped within 6 months of Screening) nicotine user, example, smokes, vapes or uses smokeless forms of tobacco such as chewing tobacco, gutka, pan containing tobacco, snus, tobacco pouches etc.
9. Participant has diagnosed xerostomia or is taking any medication or has a condition, that in the opinion of the investigator, is causing xerostomia.
10. Participant has a medical condition (example, bleeding disorder) which could directly influence gingival bleeding or could affect study outcomes and/or participant safety.
11. Participant who has a recent history (within the last year) of alcohol or other substance abuse.
12. Participant who has a severe oral condition (example, acute necrotizing ulcerative gingivitis or oral or peri-oral ulceration including herpetic lesions) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant/examiner if they participate in the study.
13. Participant has a tongue or lip piercing, or any other oral feature that, in the opinion of the investigator, could interfere with the proper usage of a toothbrush or with correct application of study products.
14. Participant has/is using the following medications:

    1. Any antibiotic medication within 28 days prior to screening, or at any time during the study.
    2. Any anti-bacterial toothpaste/mouthwash (example, chlorhexidine) or other oral care product within 2 weeks of Screening that, in the opinion of the investigator or dentally qualified designee, could affect plaque formation or gingival health.
    3. Systemic medication (example, anti-inflammatories, anticoagulants, immunosuppressants, traditional/ herbal remedy etc) within 2 weeks of screening or at any point in the study, which, in the opinion of the Investigator, could affect plaque/gingival condition (example, ibuprofen, aspirin, warfarin, cyclosporin, phenytoin, calcium channel blockers).
    4. A participant currently taking a systemic medication (example, anti-inflammatory, anticoagulant, immunosuppressants) or traditional/ herbal remedy which, in the opinion of the Investigator, could affect plaque/ gingival condition (example, ibuprofen, aspirin, warfarin, cyclosporin, phenytoin, calcium channel blockers).
15. Participant demonstrating the following dental conditions:

    1. Signs of active periodontitis (site with probing depth over 3 mm)
    2. Is receiving or has received treatment for periodontal disease (including surgery) within 12 months of Screening.
    3. Has gingivitis, which in the opinion of the investigator, is not expected to respond to treatment with an over the counter (OTC) dentifrice.
    4. Has active caries that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they participate in the study.
    5. Has dentures (partial or full) or an orthodontic appliance (bands, appliances, or fixed/ removable retainers).
    6. Has received orthodontic therapy within 3 months of Screening.
    7. Has numerous restorations in a poor state of repair.
    8. Has any dental condition (example, overcrowding) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they participate in the study.
    9. Has had dental prophylaxis or tooth bleaching within 12 weeks of Screening.
    10. Has high levels of extrinsic stain or calculus deposits, in the opinion of the investigator, that could have interfered with plaque assessments.
16. Participant who has previously been enrolled in this study.
17. Participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2025-09-09 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Mean Bleeding Index (BI) at Week 12 | Week 12
  The BI assesses the number of bleeding points elicited on probing as a measure of gingival condition. BI will be assessed on the facial and lingual gingival surfaces of each scorable tooth using a probe. The probe will be gently inserted into the gingival crevice to a depth of approximately 1 millimeter (mm) and then run around the tooth gently stretching the epithelium while sweeping from interproximal to interproximal along the sulcular epithelium. Gingival bleeding will be scored on a 3-points scale with scores ranging from 0 to 2, where 0=Absence of bleeding on probing, 1=Bleeding observed within 30 seconds of probing, 2=Bleeding observed immediately on probing. Mean BI will be calculated by taking the average over all tooth sites assessed for a participant. Lower score indicates improvement in the symptoms.

SECONDARY OUTCOMES:
Mean BI at Week 6 | Week 6
  The BI assesses the number of bleeding points elicited on probing as a measure of gingival condition. BI will be assessed on the facial and lingual gingival surfaces of each scorable tooth using a probe. The probe will be gently inserted into the gingival crevice to a depth of approximately 1 mm and then run around the tooth gently stretching the epithelium while sweeping from interproximal to interproximal along the sulcular epithelium. Gingival bleeding will be scored on a 3-points scale with scores ranging from 0 to 2, where 0=Absence of bleeding on probing, 1=Bleeding observed within 30 seconds of probing, 2=Bleeding observed immediately on probing. Mean BI will be calculated by taking the average over all tooth sites assessed for a participant. Lower score indicates improvement in the symptoms.
Mean Number of Bleeding Sites (NBS) at Weeks 6 and 12 | Week 6 and Week 12
  The NBS elicited on probing will be assessed using the BI assessment. Bleeding will be assessed on the facial and lingual gingival surfaces of each scorable tooth. The probe will be gently inserted into the gingival crevice to a depth of approximately 1 mm and then run around the tooth gently stretching the epithelium while sweeping from interproximal to interproximal along the sulcular epithelium. The NBS for each participant will be calculated as the number of tooth sites with bleeding observed immediately on probing or within 30 seconds of probing.
Mean Modified Gingival Index (MGI) at Weeks 6 and 12 | Week 6 and Week 12
  The MGI is a non-invasive assessment which focuses on the visual symptoms of gingivitis (redness, texture, edema). MGI will be assessed for all evaluable surfaces of the facial and lingual/palatal gingiva, four sites per tooth and will be scored on a 5-point scale ranging from 0 to 4, where 0 = Absence of inflammation, 1= Mild inflammation: slight change in color, little change in texture of any portion of the marginal or papillary gingival unit, 2=Mild inflammation: criteria as [1] but involving the entire marginal or papillary gingival unit, 3=Moderate inflammation: glazing, redness, edema, and/or hypertrophy of the marginal or papillary gingival unit, 4=Severe inflammation: marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration. Lower score indicates improvement in the symptoms.
Mean Overall Turesky Plaque Index (TPI) at Weeks 6 and 12 | Week 6 and Week 12
  The TPI is a non-invasive assessment of supra-gingival plaque accumulation. TPI will be assessed on the facial and lingual surfaces of each scorable tooth. Dental plaque will first be disclosed with a plaque disclosing solution and disclosed plaque will be scored using a 6-point scale ranging from 0 to 5, where 0=No plaque, 1=Separate flecks of plaque at the cervical margin, 2=Thin continuous band of plaque (up to 1 mm) at the cervical margin, 3=Band of plaque wider than 1 mm but covering less than (<) 1/3 of the tooth surface, 4=Plaque covering greater than or equal to (>=) 1/3 but < 2/3 of the tooth surface, 5=Plaque covering >= 2/3 of the tooth surface. Lower score indicates improvement in the symptoms.
Mean Interproximal TPI at Weeks 6 and 12 | Week 6 and Week 12
  The TPI is a non-invasive assessment of supra-gingival plaque accumulation. TPI will be assessed on the facial and lingual surfaces of each scorable tooth. Dental plaque will first be disclosed with a plaque disclosing solution and disclosed plaque will be scored using a 6-point scale ranging from 0 to 5, where 0=No plaque, 1=Separate flecks of plaque at the cervical margin, 2=Thin continuous band of plaque (up to 1 mm) at the cervical margin, 3=Band of plaque wider than 1 mm but covering < 1/3 of the tooth surface, 4=Plaque covering >= 1/3 but < 2/3 of the tooth surface, 5=Plaque covering >= 2/3 of the tooth surface. Lower score indicates improvement in the symptoms.
Change from Baseline in Salivary Tin Concentration Pre- and Post-brushing at Weeks 6 and 12 | Baseline, Week 6 and Week 12: Pre-brushing and at 15, 30, 60, 120 minutes post-brushing
  Unstimulated saliva samples will be collected from participants pre- and post-brushing. The samples will be analyzed for tin concentration to investigate the retention of the stannous [tin(II)] ion within the oral cavity. Change from baseline in salivary tin concentration at indicated timepoints will be reported.
Area Under the Curve (AUC) of Salivary Tin Concentration Post-brushing at Baseline, Weeks 6 and 12 | Baseline, Week 6 and Week 12: Pre-brushing and at 15, 30, 60, 120 minutes post-brushing
  Unstimulated saliva samples will be collected from participants pre- and post-brushing for the analysis of salivary tin concentration. The AUC [pre-treatment, t=0 to 120 minutes] values for the change from baseline in the log10 transformed salivary tin concentrations versus (vs) time will be reported.
Salivary Tin Concentration Pre-brushing at Baseline, Weeks 6 and 12 | Baseline, Week 6 and Week 12
  Unstimulated saliva samples will be collected from participants pre- and post-brushing. The samples will be analyzed for tin concentration to investigate the retention of the stannous [tin(II)] ion within the oral cavity. Salivary tin concentration at the indicated timepoints will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- All Sum Research, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.